CLINICAL TRIAL: NCT04217915
Title: A Survey of Management of Analgesia, Sedation and Delirium in ICU Patients in China
Acronym: SASE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Peking University People's Hospital (Other); Qilu Hospital of Shandong University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Jilin University (Other); General Hospital of Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Xiaochun Ma,MD, director of ICUof first hospital of China medical university, China Medical University, China
Other Study IDs: CMU1h
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Delirium on Emergence; Analgesia; Separation
Keywords: analgesia; sedation; ICU; Delirium
MeSH Terms: conditions — Emergence Delirium; Agnosia; Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2018, the severe medicine branch of the Chinese Medical Association and the American Society of severe medicine successively updated the pain and sedation guidelines for severe patients (PADIS guidelines). In addition to the update of the original evaluation and management of pain and sedation and delirium, the new guidelines also increased the monitoring and management of early activities and sleep quality for severe patients. Therefore, it is necessary for us to investigate the compliance of the new guidelines for analgesia, sedation and delirium management among the medical staff of critical care, so as to find out the existing problems in the management of analgesia, sedation and delirium in critical care patients, and find solutions to improve the overall quality level of our management of critical care patients

DETAILED DESCRIPTION:
The first part is to master the current situation of analgesia, sedation and delirium management of ICU patients in China. In order to understand the compliance of Chinese ICU doctors and nurses with the PADIS guidelines, a questionnaire survey was conducted with the participation of multiple centers in China, aiming at the doctors and nurses with different seniority in the critical medicine department. At the same time, the total number of critically ill patients, pain, agitation and delirium assessment tools and critical patients in 2018 were investigated The incidence of pain, agitation and delirium, the implementation of early activities, the monitoring and evaluation of sleep quality, and related interventions, including real-world clinical data such as drug treatment and non drug treatment.The second part focuses on the management of severe delirium in ICU in China. For the patients with delirium in the above survey, a further in-depth and detailed survey shall be conducted, covering the basic diseases of the patients, the occurrence time of delirium, the type of delirium, relevant risk factors, the diagnosis method of delirium, the duration of delirium, the prevention and treatment measures (including drug treatment and non drug treatment measures), and the prognosis of delirium patients .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* stay in ICU for more than 24 hours and have used analgesics and Sedatives.

Exclusion Criteria:

* Before entering the ICU, they had mental illness and dementia;
* coma or deep sedation could not be evaluated;
* brain injury, stroke sequelae, epilepsy and other brain diseases;
* nerious audio-visual dysfunction and unable to communicate normally.
* Pregnant and lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were randomly selected from the ICU of the A tertiary hospitals in the major provinces and cities of China.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-07-12 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance of ICU medical staff with PADIS guidelines | 2020.12
  The assessment tool is a self-designed questionnaire based on the guidelines, which is mainly used to assess the compliance of medical staff with the guidelines in their daily work

SECONDARY OUTCOMES:
Incidence of delirium | 2020.12
  Incidence of delirium in Chinese ICU patients with analgesia and sedation during the study period

CONTACTS AND LOCATIONS:
Overall Officials: xiaochun ma, doctor, Study Chair — China Medical University, China
Locations (1):
- the first hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang J, Peng ZY, Zhou WH, Hu B, Rao X, Li JG. A National Multicenter Survey on Management of Pain, Agitation, and Delirium in Intensive Care Units in China. Chin Med J (Engl). 2017 May 20;130(10):1182-1188. doi: 10.4103/0366-6999.205852. PMID 28485318
- [Result] Morandi A, Piva S, Ely EW, Myatra SN, Salluh JIF, Amare D, Azoulay E, Bellelli G, Csomos A, Fan E, Fagoni N, Girard TD, Heras La Calle G, Inoue S, Lim CM, Kaps R, Kotfis K, Koh Y, Misango D, Pandharipande PP, Permpikul C, Cheng Tan C, Wang DX, Sharshar T, Shehabi Y, Skrobik Y, Singh JM, Slooter A, Smith M, Tsuruta R, Latronico N. Worldwide Survey of the "Assessing Pain, Both Spontaneous Awakening and Breathing Trials, Choice of Drugs, Delirium Monitoring/Management, Early Exercise/Mobility, and Family Empowerment" (ABCDEF) Bundle. Crit Care Med. 2017 Nov;45(11):e1111-e1122. doi: 10.1097/CCM.0000000000002640. PMID 28787293